CLINICAL TRIAL: NCT04049864
Title: Pilot Clinical Study of DNA Vaccination Against Neuroblastoma
Brief Title: DNA Vaccination Against Neuroblastoma
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Belarusian Research Center for Pediatric Oncology, Hematology and Immunology (Other)
Responsible Party: Principal Investigator, Alexander Meleshko, Principal Investigator, Belarusian Research Center for Pediatric Oncology, Hematology and Immunology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BelarusianPediatric
Record Dates: First submitted 2019-07-31; First posted 2019-08-08 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Relapsed Neuroblastoma
Keywords: neuroblastoma; DNA vaccine; Salmonella vaccine; polyethylenimine
MeSH Terms: conditions — Neuroblastoma | interventions — Vaccines, DNA; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All subjects (Experimental): All subjects will receive the vaccine and be followed per the schedule of procedures.
  Interventions: Biological: DNA vaccine; Biological: Salmonella oral vaccine; Drug: Lenalidomide

INTERVENTIONS:
Biological: DNA vaccine — conjugate of plasmid DNA with linear polyethylenimine 20 kDa (PEI) One dose includes 400 µg of DNA and 500 µg of PEI.
  Other Names: DNA-PEI polyplex
Biological: Salmonella oral vaccine — suspension 10^10 CFU of an attenuated Salmonella enterica serovar typhimurium strain (SS2017) containing the plasmid of the corresponding DNA vaccine.
Drug: Lenalidomide — Lenalidomide is prescribed in a dose of 25 mg / day in a course of three weeks starting 7 days before the first vaccination course and ending on the day of the last vaccination course.

SUMMARY:
This is pilot open-label study to evaluate the safety and immunogenicity of a DNA vaccine strategy in relapsed neuroblastoma patients following chemotherapy and HSC transplantation. The combined form of the vaccine includes an intramuscular injection of the DNA-polyethylenimine conjugate and oral administration using the attenuated Salmonella enterica as DNA vaccine carriers.

Objectives of the study:

1. To assess safety and document local and systemic toxicity to combined DNA vaccine
2. To determine immunogenicity of the vaccine
3. To evaluate clinical response to vaccination. Control of minimal residual disease in bone marrow and duration of remission.

DETAILED DESCRIPTION:
DNA vaccine construction includes chimeric fusion of neuroblastoma-associated antigen and potato virus X coat protein (PVXCP) as an immune enhancer. In each course vaccine for one antigen is applies. The selection of antigens is carried out after analyzing of their expression in the tumor biopsy material by PCR and IHC. The list of antigens used in the study: tyrosine hydroxylase (TH), Phox2B, Survivin, MAGEA1, MAGEA3, PRAME. The antigens with the highest level of expression in the tumor sample of each patient are selected for vaccination.

Vaccination schedule for each patient includes three courses of vaccination. One course includes three administrations of vaccines against a single antigen. Vaccination is repeated at intervals of 1 week (plus minus 3 working days). Break between courses - 3-4 weeks. Each vaccination includes an injection and taking a capsule with a dose of bacteria.

For intramuscular injection, we use conjugate (polyplex) DNA with linear polyethylenimine 20 kDa (PEI). One dose includes 400 µg of DNA and 500 µg of PEI. When administered orally, the patient receives a suspension 10^10 CFU of an attenuated Salmonella enterica serovar typhimurium strain (SS2017) containing the plasmid of the corresponding DNA vaccine.

Before and during vaccination, an accompanying chemotherapy is carried out, including cyclophosphamide, propranolol, celecoxib and lenalidomide. Cyclophosphamide is prescribed three days before the start of each vaccination course in a single dose of 300 mg / m2. Lenalidomide is prescribed in a dose of 25 mg / day in a course of three weeks starting 7 days before the first vaccination course and ending on the day of the last vaccination course

ELIGIBILITY:
Inclusion Criteria:

1. The diagnosis of neuroblastoma recurrence with morphological / cytological confirmation;
2. The presence of tumor tissue for biopsy;
3. The absence of progression or a large tumor mass (bulky disease);
4. The physical status on the scale of ECOG 0 - 2.
5. Life expectancy of at least 12 months
6. Indicators of cellular immunity of the blood: lymphocytes - at least 1 * 10^9;
7. Availability of written informed consent of the patient and his parents (legal representatives) to participate in this protocol.
8. Compliance of parents (legal representatives) and the patient himself with participation in the study protocol.

Exclusion Criteria:

A. Based on the anamnesis:

1. The presence of any primary immunodeficiency;
2. The presence of a primary multiple malignant tumor;
3. The presence of autoimmune diseases in history (except thyroiditis);
4. Polyalgia;
5. Severe diseases, including those with severe symptoms, untreated inflammatory and infectious processes, due to which the patient cannot receive treatment in accordance with the study protocol.
6. Socioeconomic or geographical circumstances that cannot guarantee proper compliance with the requirements of the protocol for treatment and further observation.

B. based on survey data:

1. The absence of expression in the tumor tissue of two or more antigens used in the protocol;
2. The level of peripheral blood leukocytes <1.5 × 10^9 /L, platelet <50.0 × 10^9 /L, Hemoglobin less than 80 g / L;
3. Positive tests for human immunodeficiency virus (HIV), hepatitis B or C.
4. Severe impaired liver function - the levels of AST / SGOT or ALT / SGPT exceed the upper limit of normal 5 times or more.

Ages: 1 Year to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-01-09 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events experienced by subjects | for 3 months from the first vaccination
  To assess the safety of the DNA-PEI and Salmonella vaccines
Immune response to the vaccine | In check point after 2nd course (9 week after first vaccine)
  Immunogenicity will be evaluated by assessing T-cell IFN-γ production in ELISPOT and PVXCP antibody production by ELISA
Immune response to the vaccine | In check point after 3rd course (14 week after the first vaccine)
  Immunogenicity will be evaluated by assessing T-cell IFN-γ production in ELISPOT and PVXCP antibody production by ELISA
Minimal residual disease - MRD | up to 4 weeks after the last vaccination
  MRD in bone marrow measured by RQ-PCR and flow cytometry

SECONDARY OUTCOMES:
Progression free survival - PFS | Up to 12 months
  Time from treatment to date of first documented progression or date of death

CONTACTS AND LOCATIONS:
Overall Officials: Inna V Proleskovskaya, PhD, MD, Study Director — Belarussian Research Center for Pediatric Oncology, Hematology and Immunology
Locations (1):
- Belarussian Research Center for Pediatric Oncology, Hematology and Immunology, Minsk, Minsk Oblast, Belarus